CLINICAL TRIAL: NCT05663177
Title: Almonertinib Plus Metronomic Oral Vinorelbine Beyond Limited Progression on Third-generation TKI in EGFR-mutant Advanced NSCLC，an Observational Study
Brief Title: Almonertinib Plus Metronomic Oral Vinorelbine
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: SCOG005
Record Dates: First submitted 2022-12-06; First posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: EGFR; NSCLC; Third-generation TKI
MeSH Terms: interventions — aumolertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Study arm: Almonertinib plus metronomic oral vinorelbine
  Interventions: Drug: Almonertinib and metronomic oral vinorelbine

INTERVENTIONS:
Drug: Almonertinib and metronomic oral vinorelbine — Ametinib 110mg once a day; Oral Vinorelbine 40mg three times a week for three weeks and Q28d for one course.

SUMMARY:
To evaluate the efficacy of continuing osimertinib in conjunction with metronomic oral vinorelbine after limited progression on osimertinib, to provide clinical experience on the treatment strategy for these patients.

DETAILED DESCRIPTION:
This study is a clinical observation study. The patients who comfirm the criteria will be treated with Almonertinib plus metronomic oral vinorelbine. The patients will be followed up until the tumor progressed, and the efficacy (PFS, ORR, DCR) of tumor therapy were evaluated.

Drug administration regimen: Ametinib 110mg once a day; Oral Vinorelbine 40mg three times a week for three weeks and Q28d for one course.

ELIGIBILITY:
Inclusion Criteria:

* Non-small cell lung cancer diagnosed by histopathology or cytology;
* Previous molecular pathology was EGFR sensitive mutation;
* Stage IV;
* ECOG score 0-2;
* Prior to receiving the third generation of EGFR-TKI targeted therapy, and TKI targeted therapy showed limited progress;
* According to RECIST1.1 standards, there are measurable or evaluable lesions
* The patient has fully understood this study and voluntarily signed a written informed consent form;
* The estimated survival time is more than 3 months.

Exclusion Criteria:

* Histological or cytological confirmation of small cell lung cancer or squamous cell carcinoma at the first diagnosis;
* The progression of the third generation EGFR-TKI suggests histological transformation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EGFR-mutant advanced NSCLC, disease progression on the third-generation TKI
Sampling Method: Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2022-12-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 100 months
  progression-free survival

SECONDARY OUTCOMES:
ORR | up to 12 months
  Objective Response Rate
DCR | up to 12 months
  Disease Control Rate

IPD SHARING:
Plan to Share IPD: No